CLINICAL TRIAL: NCT05059041
Title: Dilated Wavefront Versus Non-Dilated Wavefront for Metric-Optimized Refraction Procedure for Individuals With Down Syndrome
Brief Title: Dilated Versus Non-Dilated Wavefront Corrections for Patients With Down Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Heather Anderson OD, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EY024590
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Down Syndrome; Refractive Errors
MeSH Terms: conditions — Down Syndrome; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dilated first, non-dilated second (Experimental): Each participant will perform vision testing first through a prescription determined from wavefront measurements obtained after dilation. Second, each participation will perform vision testing through a prescription determined from wavefront measurements obtained before dilation.
  Interventions: Device: Dilated Refraction; Device: Non-Dilated Refraction
- Non-dilated first, dilated second (Experimental): Each participant will perform vision testing first through a prescription determined from wavefront measurements obtained before dilation. Second, each participation will perform vision testing through a prescription determined from wavefront measurements obtained after dilation.
  Interventions: Device: Dilated Refraction; Device: Non-Dilated Refraction

INTERVENTIONS:
Device: Dilated Refraction — The dilated refraction will be a trial spectacle frame composed of lenses based upon a spectacle prescription determined from dilated measures of the eye using a wavefront aberrometer.
Device: Non-Dilated Refraction — The non-dilated refraction will be a trial spectacle frame composed of lenses based upon a spectacle prescription determined from non-dilated measures of the eye using a wavefront aberrometer.

SUMMARY:
Individuals with Down syndrome (DS) live with visual deficits due, in part, to elevated levels of higher-order optical aberrations (HOA). HOAs are distortions/abnormalities in the structure of the refractive components of the eye (i.e. the cornea and the lens) that, if present, can result in poor quality focus on the retina, thus negatively impacting vision. HOAs in the general population are overall low, and thus not ordinarily considered during the eye examination and determination of refractive correction. However, for some populations, such as individuals with DS, HOAs are elevated, and thus the commonly used clinical techniques to determine refractive corrections may fall short. The most common clinical technique for refractive correction determination is subjective refraction whereby a clinician asks the patient to compare different lens options and select the lens that provides the best visual outcome. Given the cognitive demands of the standard subjective refraction technique, clinicians rely on objective clinical techniques to prescribe optical corrections for individuals with DS. This is problematic, because it may result in errors for eyes with elevated HOA given that these techniques do not include measurement of the HOAs. The proposed research evaluates the use of objective wavefront measurements that quantify the HOAs of the eye as a basis for refractive correction determination for patients with DS. The specific aim is to determine whether dilation of the eyes is needed prior to objective wavefront measurements. Dilation of the eyes increases the ability to measure the optical quality of the eye and paralyzes accommodation (the natural focusing mechanism of the eye), which could be beneficial in determining refractions. However, the use of dilation lengthens the process for determining prescriptions and may be less desirable for patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* Able to be dilated
* Able to fixate for study measures
* Able to respond for visual acuity testing

Exclusion Criteria:

* Ocular nystagmus
* History of ocular or refractive surgery (strabismus surgery is okay)
* Corneal or lenticular opacities
* Ocular disease

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Distance Visual Acuity | 1 day
  Distance LogMAR visual acuity will be measured with the British Standard Letter set or HOTV Matching for participants unable to name letters

SECONDARY OUTCOMES:
Near Visual Acuity | 1 day
  Near LogMAR visual acuity will be measured with a Bailey-Lovie style HOTV card.
Participant distance vision ranking | 1 day
  Participants will be asked rate quality of vision at distance on a five point scale for each prescription. 1 will correspond to poorest vision and 5 will correspond to best vision.
Participant near vision ranking | 1 day
  Participants will be asked rate quality of vision at near on a five point scale for each prescription. 1 will correspond to poorest vision and 5 will correspond to best vision.
Participant overall preference for prescriptions | 1 day
  Participants will be asked to select which of two prescriptions are preferred overall.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Anderson, OD, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - University of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided